CLINICAL TRIAL: NCT04826484
Title: A Randomized Trial Evaluating Use of Long-Acting Liposomal Bupivacaine (Exparel®) in Reducing Narcotic Pain Requirements in Pediatric Patients Undergoing Minor Urologic Procedures
Brief Title: Opioid Reduction Initiative During Outpatient Pediatric Urologic Procedures Using Exparel
Acronym: Baby ORIOLES
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Met futility threshold at interim analysis
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00284462
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Urologic Diseases; Hypospadias; Undescended Testes; Chordee; Hydrocele; Orchiectomy
MeSH Terms: conditions — Urologic Diseases; Hypospadias; Cryptorchidism; Testicular Hydrocele | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivacaine plus 0.25% Bupivacaine (Experimental): Participants will receive local wound infiltration with sequential Liposomal Bupivacaine plus 0.25% Bupivacaine
  Interventions: Drug: Exparel 133 miligrams per 10 milliliter injection; Drug: Bupivacaine Hydrochloride
- 0.25% Bupivacaine alone (Active Comparator): Participants will receive local wound infiltration with 0.25% Bupivacaine alone.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Exparel 133 miligrams per 10 milliliter injection — Local wound infiltration with Exparel 133 miligrams per 10 milliliter injection
  Arms: Liposomal Bupivacaine plus 0.25% Bupivacaine
Drug: Bupivacaine Hydrochloride — Local wound infiltration with 0.25% bupivacaine.

SUMMARY:
This study aims to evaluate the utility of long-acting liposomal bupivacaine (Exparel®) in improving pain scores and reducing narcotic pain requirements in pediatric patients following minor urologic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients 6 years and older undergoing minor pediatric urologic surgery
* Patients who are otherwise eligible to receive routine care following minor urologic surgery

Exclusion Criteria:

* Contraindication to receiving local anesthetics (i.e. pre-existing cardiac, renal, hepatic dysfunction)
* Pediatric patients younger than 6 years of age
* Pediatric patients with a history of pain syndromes or are unable to tolerate opiate medication
* Unwilling to participate in 48 hours and 10-14 day follow-up phone calls

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather N DiCarlo, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gabrielson AT, Galansky L, Sholklapper T, Crigger C, Patel HD, Harris K, Haney N, Jing Y, Wang MH, Wu C, Gearhart JP, Di Carlo HN. Effectiveness of Liposomal Bupivacaine With Bupivacaine Hydrochloride vs Bupivacaine Hydrochloride Alone as a Local Anesthetic for Children Undergoing Ambulatory Urologic Surgery: The Baby ORIOLES Randomized Clinical Trial. J Urol. 2024 Jan;211(1):37-47. doi: 10.1097/JU.0000000000003764. Epub 2023 Oct 23. PMID 37871332

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine Plus 0.25% Bupivacaine | 0.25% Bupivacaine Alone
Started | 52 | 52
Completed | 50 | 52
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine Plus 0.25% Bupivacaine | 0.25% Bupivacaine Alone | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 9.5 [8 to 13] | 11 [8 to 12] | 10 [8 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 52 | 52 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 29 | 32 | 61
  Race: African American | 13 | 7 | 20
  Race: Asian | 5 | 9 | 14
  Race: LatinX/Hispanic | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 52 | 104
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 18.5 [16 to 21] | 18.6 [16 to 20] | 18.5 [16 to 20]
Procedure Type [Count of Participants; unit: Participants]
  Orchiopexy | 20 | 21 | 41
  Circumcision | 20 | 22 | 42
  Distal Hypospadias Repair | 0 | 1 | 1
  Inguinal Hernia Repair/Hydrocelectomy | 5 | 7 | 12
  Penile Cyst Excision | 1 | 0 | 1
  Chordee Repair | 6 | 1 | 7
Postoperative Pain Management Strategies [Number; unit: participants]
  Ketoralac | 30 | 38 | 68
  Tylenol | 48 | 47 | 95
  Ibuprofen plus Tylenol | 32 | 29 | 61
Surgeon Performing Procedure [Count of Participants; unit: Participants]
  Surgeon 1 | 14 | 9 | 23
  Surgeon 2 | 7 | 17 | 24
  Surgeon 3 | 9 | 11 | 20
  Surgeon 4 | 22 | 15 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Are Opiate-free
Description: Percentage of patients who are opiate-free at 48 hours postoperatively.
Time Frame: 48 hours postoperatively
Measure: Number; unit: percentage of patients opioid-free
Arm/Group | Liposomal Bupivacaine Plus 0.25% Bupivacaine | 0.25% Bupivacaine Alone
Number analyzed (Participants) | 52 | 52
percentage of patients opioid-free | 60 | 62

2. Primary Outcome: Percentage of Patients Who Are Opiate-free at 10-14 Days Postoperatively
Description: Percentage of patients who are opiate-free at 10-14 days postoperatively.
Time Frame: 10-14 days postoperatively
Population: Two patients in the intervention arm were lost to follow-up at the 10-14d followup (thus 50 were available for analysis)
Measure: Number; unit: percentage of pt opioid-free at 10-14d
Arm/Group | Liposomal Bupivacaine Plus 0.25% Bupivacaine | 0.25% Bupivacaine Alone
Number analyzed (Participants) | 50 | 52
percentage of pt opioid-free at 10-14d | 60 | 62

3. Primary Outcome: Parents' Postoperative Pain Measure (PPPM) Scores
Description: 15-item, yes/no behavioral checklist based on non-verbal pain cues children show following surgery. Scale is from 0 to 15, with higher scores denoting more severe pain. A score of 6+ has been validated as a threshold for a child experiencing clinically significant pain.
Time Frame: 48 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine Plus 0.25% Bupivacaine | 0.25% Bupivacaine Alone
Number analyzed (Participants) | 52 | 52
score on a scale | 2 [1 to 3] | 2.5 [2 to 4]

4. Primary Outcome: Parents' Postoperative Pain Measure (PPPM) Scores
Description: as for outcome 3
Time Frame: 10-14 days postoperatively
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine Plus 0.25% Bupivacaine | 0.25% Bupivacaine Alone
Number analyzed (Participants) | 50 | 52
score on a scale | 0 [0 to 1] | 0 [0 to 1]

5. Secondary Outcome: Amount of Opioid Medication Used Post-discharge
Description: Weight based amount of opioid medication (in OMEQ/kg) used post-discharge.
Time Frame: 10-14 days postoperatively
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Oral morphine equivalent per kg (OMEQ/kg
Arm/Group | Liposomal Bupivacaine Plus 0.25% Bupivacaine | 0.25% Bupivacaine Alone
Number analyzed (Participants) | 50 | 52
Oral morphine equivalent per kg (OMEQ/kg | 0 [0 to 0.1] | 0 [0 to 0.22]

6. Secondary Outcome: Percentage of Patients With Leftover Opioid Medication
Description: Percentage of patients with leftover opioid medication
Time Frame: 10-14 days postoperatively
Population: as for outcome 2
Measure: Number; unit: % of patients with leftover opiates
Arm/Group | Liposomal Bupivacaine Plus 0.25% Bupivacaine | 0.25% Bupivacaine Alone
Number analyzed (Participants) | 50 | 52
% of patients with leftover opiates | 14 | 24

7. Secondary Outcome: Cumulative Incidence of Complications Related to Local Anesthetic Systemic Toxicity
Description: Cumulative incidence of complications related to local anesthetic systemic toxicity
Time Frame: 10-14 days postoperatively
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine Plus 0.25% Bupivacaine | 0.25% Bupivacaine Alone
Number analyzed (Participants) | 50 | 52
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Liposomal Bupivacaine Plus 0.25% Bupivacaine | 0.25% Bupivacaine Alone
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 7/52 | 5/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Bupivacaine Plus 0.25% Bupivacaine (N=52) | 0.25% Bupivacaine Alone (N=52)
Postoperative swelling (Renal and urinary disorders) | 6 (6) | 5 (5) — Postoperative swelling prompting a phone call/message to the office
Penile Hematoma (Renal and urinary disorders) | 1 (1) | 0 (0) — Hematoma

LIMITATIONS AND CAVEATS:
The trial met the predetermined threshold for early stopping.

1. Inability to blind surgeons due to differences in the appearance of the agents.
2. Unclear if the absorption profile of intervention is more rapid in groin/dorsal penile tissue compared to other areas.
3. Our cohort was enriched with low morbidity procedures which may have decreased differences between arms
4. Inability to compare the efficacy of the agents stratified by procedure type due to low enrollment in each procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT04826484/Prot_SAP_000.pdf